CLINICAL TRIAL: NCT04765917
Title: Effect of Motor Imagery Training on Gait and Balance in Children With Spastic Hemiplegia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Eman Kamal Abdelmoteleb, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Ekamal_phd2021
Record Dates: First submitted 2021-02-16; First posted 2021-02-23 (Actual); Last update posted 2021-04-13 (Actual); Status verified 2021-04

CONDITIONS: Cerebral Palsy, Spastic
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Intervention Model Description: 2 different groups receive different interventions at the same time during the study
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Selected Physical Therapy group (Active Comparator): The Control group will receive a selected physical therapy program for 60 minutes, 3 times/week for 3 successive months including the following exercises
  Interventions: Other: Selected physical Therapy program
- Motor imagery training (Experimental): Children allocated to the study group will receive the same selected physical therapy program given to the control group for 30 min in addition to 30 minutes motor imagery training program
  Interventions: Other: Selected physical Therapy program; Other: Motor imagery training program

INTERVENTIONS:
Other: Selected physical Therapy program — -Facilitation of balance reactions from standing position including: Standing on one leg, weight shifting from standing position, stoop and recover from standing, squat from standing, standing on balance board and pushing the child in different directions.
  * Facilitation of counterpoising mechanism through instructing the child to kick ball from standing position as well as catching and throwing ball with his hands.
  * Strengthening exercises for weakened muscles in upper and lower limbs muscle.
  * Strengthening exercises for back and abdominal muscles.
  * Stretching exercises for tight muscles in upper and lower limbs.
  * Gait training activities for correction of gait pattern including: walking on balance beam, walking on balance board, walking on uneven surface, walking using different obstacles (rolls, wedges, stepper) and walking up and down stairs.
  * Jumping in place and jumping a board.
Other: Motor imagery training program — As a preparation each child will be shown a video of 5 minutes of normal movements.
  They will be positioned in a comfortable position. The screen is in the child's visual field. Children will be asked to close their eyes and imagine they will perform the physically practiced task for 10 minutes, similar to one shown in the video. Sequence of the task will be verbally explained to the child for better recalling of sensations in muscles during the movements. During the entire exercise schedule child's attention will be focused on the position, and movement of their body, on proprioceptive inputs coming from the leg muscles and on the tactile sensations of foot floor contact.
  Thereafter, the child will be asked to perform the sequence of tasks, rehearsed mentally for 20 minutes.
  Arms: Motor imagery training

SUMMARY:
This study aims to:

* Investigate the effect of motor imagery training on gait kinematics in children with spastic hemiplegia.
* Determine the effect of motor imagery training on balance in children with spastic hemiplegia.
* Assess the effect of motor imagery training on trunk endurance in children with spastic hemiplegia.

DETAILED DESCRIPTION:
Children with spastic hemiplegia may experience a variety of concomitant health conditions including, movement difficulty, postural and balance instability, muscle spasticity, difficulty with motor planning and control, and cognitive impairments.

Postural and balance disturbances occur due to the difficulty in maintaining the body segments aligned on narrow base of support and there is limitation in balance recovery in hemiplegic children contributing to delayed responses of ankle muscles, inappropriate sequencing, and increased coactivation of agonists/ antagonists muscles.

Treatment will vary depending on the severity of impairments, level of activity, participation, and on the priorities highlighted by the patient. Walking is often identified as a main goal, and there is evidence that children with hemiplegia can take steps before regaining standing balance, which would support early walking. Many advanced treatment approaches are used to help improve motor function and gait in patients with hemiplegic CP.

Rehabilitation techniques are predominantly focused on alleviating the compromised motor execution facet of action performance, and have not specifically targeted the motor preparation or planning processes. Motor imagery is proposed to be a backdoor mechanism to access the motor system. It being a theoretically feasible method to activate the immature networks involved in motor control. Therefore, for individuals with motor planning problems this cognitive MI training may be useful to improve motor skills.

Although it has been shown to be beneficial in adult patients with stroke, and it still awaits empirical testing in young children with CP.

Despite the potential benefits of motor imagery training, clinical use of motor imagery training for improving walking and balance abilities is not yet common compared with other conventional modalities in rehabilitation of children with hemiplegia. Consequently, more research and further confirmation are needed regarding the impact of motor imagery training on the gait performance, balance and trunk endurance in children with hemiplegia. Therefore, the purpose of this study to investigate the effect of motor imagery training on balance and kinematic parameters of gait in children with hemiplegia.

ELIGIBILITY:
Inclusion Criteria:

* Their chronological age will be ranged from 7-10 years.
* Their motor function will be at level I according to according to Gross Motor Function Classification System GMFCS (Palisano et al., 2008).
* The degree of spasticity for these children will ranged from grade 1 to 1+ according to Modified Ashworth Scale (Bohannon and Smith, 1987).
* They will be able to follow instructions during evaluation and treatment.

Exclusion Criteria:

Children will be excluded from the study if they have:

* Cardiovascular or respiratory disorders.
* Botulinium muscular injection in the last 6 months
* Surgical interference in lower limbs.
* Musculoskeletal problems or fixed deformities in the spine and/or lower extremities.
* Seizures.
* Visual or hearing impairment.
* Mentally retarded children

Ages: 7 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2021-02-01 (Actual); Primary Completion 2022-03-01 (Estimated); Study Completion 2022-04-01 (Estimated)

PRIMARY OUTCOMES:
Assessing the change in Spatial parameters of gait | "through study completion, an average of 3 months"
  Analysis of Spatial parameters of gait by using Kinovea software via 2D gait analysis in order to measure the changes in: stride length (cm), Step length (cm).
Assessing the change in cadence | "through study completion, an average of 3 months"
  Analysis of temporal parameters of gait by using Kinovea software via 2D gait analysis in order to measure the changes in: cadence (number of steps / minute).
Assessing the change in Angular displacement of joint in gait cycle | "through study completion, an average of 3 months"
  Analysis of Angular displacement of joint in gait cycle by using Kinovea software via 2D gait analysis in order to measure the changes in: Ankle dorsiflexion angle in initial contact, hip flexion angle at initial swing and knee extension at midstance. All of these parameters will be measured in degrees.
Assessing the change in Balance | "through study completion, an average of 3 months"
  Evaluation of balance by using HUMAC balance system in order to measure the change in: modified clinical test of sensory integration test (score), limits of stability (score) and weight shift (score). The highest score is (100) and the lower score is (0). The higher scores means a better outcome.
Assessing the change in walking speed | "through study completion, an average of 3 months"
  Analysis of temporal parameters of gait by using Kinovea software via 2D gait analysis in order to measure the changes in: walking speed (meter / minute).

SECONDARY OUTCOMES:
Assessing the change in Trunk muscles endurance | "through study completion, an average of 3 months"
  Evaluation of trunk muscles endurance by using 3 isometric endurance tests in order to measure the change in trunk muscle endurance via using: Trunk flexion endurance test (seconds), trunk extension endurance test (seconds) and lateral trunk endurance test (seconds)

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Physical Therapy - Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided